CLINICAL TRIAL: NCT00723463
Title: Retrospective - Prospective - Study to Determine if Apparent Diffusion Coefficient (ADC) Values Can Differentiate Tumors From Normal Tissues at 3T MRI
Brief Title: Determine if Apparent Diffusion Coefficient (ADC) Values Can Differentiate Tumors From Normal Tissue
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Ashok Srinivasan, M.D., Principal Investigator, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HUM 5527
Record Dates: First submitted 2008-07-24; First posted 2008-07-28 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Brain Cancer; Neck Cancer
MeSH Terms: conditions — Brain Neoplasms; Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): To determine if apparent diffusion coefficient values can differentiate tumors from normal tissues using a 3T MRI scan.
  Interventions: Procedure: 3T MRI scan

INTERVENTIONS:
Procedure: 3T MRI scan — Establishing/evaluating apparent diffusion coefficient (ADC) values using a 3T MRI scan to differentiate tumors from normal tissue.

SUMMARY:
The purpose of this study is to determine normal measurements (ADC values) from the head and neck of healthy volunteers using 3T MRI.

DETAILED DESCRIPTION:
The purpose of this study is to determine normal measurements (ADC values) from the head and necks of healthy subjects using 3T MRI.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects 18 years of age or older.

Exclusion Criteria:

* Under 18 years of age
* Women of child bearing potential
* Pregnant or lactating women
* All potential volunteers will be pre-screened by MRI personnel to determine if there is any medical reason that you should not be included in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2006-06; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
To determine if ADC values determined at 3T are different between normal tissues and tumors arising from the extracranial head and neck. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ashok Srinivasan, M.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Health System, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No